CLINICAL TRIAL: NCT05403866
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Multiple Doses of LT3001 Drug Product in Subjects With Acute Ischemic Stroke (AIS)
Brief Title: A Study to Evaluate the Safety and Efficacy of Multiple Doses of LT3001 Drug Product in AIS Subjects
Acronym: BRIGHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lumosa Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LT3001-205
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Results first posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LT3001 Drug Product (Experimental): Administered by intravenous infusion
  Interventions: Drug: LT3001 Drug Product
- Placebo (Placebo Comparator): Administered by intravenous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LT3001 Drug Product — Administered by intravenous infusion
  Arms: LT3001 Drug Product
Drug: Placebo — Administered by intravenous infusion
  Arms: Placebo

SUMMARY:
This is a phase II, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of multiple doses of LT3001 drug product in subjects with acute ischemic stroke (AIS)

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, and placebo-controlled prospective Phase II clinical study, designed to evaluate LT3001 drug product versus placebo in subjects with AIS. The study is planned to take place in multiple countries. Subjects who participate in this trial should be treated with standard of care of AIS therapies when appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18 to 90 years.
2. Subject has an NIHSS of 6 to 25.
3. Subject is able to receive the first IP within 24 hours after stroke symptoms onset.

Neuroimaging Inclusion Criteria:

1. Subject is able to undergo a contrast brain perfusion with either MRI or computed tomography (CT).
2. Subject has Target Mismatch Profile on MRI (perfusion is included) or CTP: ischemic core volume ≤70 mL, mismatch ratio ≥1.2 and mismatch volume ≥5 mL.

Exclusion Criteria:

1. Subject has been treated or intent to treat with endovascular thrombectomy and/or intravenous thrombolytic during the current AIS.
2. Subject has a pre-stroke disability (mRS ≥2).
3. Subject has large ischemic core volume >70 mL or ASPECTS ≤5.
4. Subject has symptoms of suspected subarachnoid hemorrhage.
5. Subject has imaging evidence of acute intracranial hemorrhage, intracranial tumor, arteriovenous malformations, other central nervous system lesions that could increase the risk of bleeding, or aneurysm requiring treatment.
6. Subject has significant mass effect with midline shift.
7. Subject has pre-existing medical, neurological, or psychiatric disease that would confound the neurological or functional evaluations.
8. Subject has current uncontrolled hypertension despite treatment.
9. Subject has INR >1.7 or abnormal aPTT or platelet count <100,000/mm^3.
10. Subject has received conventional heparin or new oral anticoagulants within 48 hours before the first IP administration.
11. Subject has blood glucose concentration <50 mg/dL or >400 mg/dL.
12. Subject has moderate or severe hepatic, renal, and/or active infectious disease.
13. Subject is lactating, pregnant, or planning to become pregnant during the study.
14. Subject has had history of sICH, prior AIS, myocardial infarction, or serious head trauma within 90 days before Screening.
15. Subject has had any major surgery within 90 days before Screening.
16. Subject has had a bleeding event within 21 days before Screening.
17. Subject has puncture of noncompressible vessels within 7 days before Screening.
18. Subject has participated in another investigational study and received IP within 30 days before Screening or 5 half-lives (whichever is longer).
19. In the opinion of the Investigator, the subject is not appropriate for the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chattanooga Center for Neurologic Research, Chattanooga, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LT3001 Drug Product | Placebo
Started | 43 | 45
Completed | 37 | 42
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | LT3001 Drug Product | Placebo | Total
Number analyzed (Participants) | 43 | 45 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (12.28) | 65.7 (11.38) | 66.5 (11.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 29 | 32 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 22 | 20 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 18 | 23 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Weight [Mean (Standard Deviation); unit: Kg] | 74.75 (16.723) | 74.28 (17.827) | 74.51 (17.198)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects With Adverse Events (AEs), Judged to be Probably or Definitely Related to the Investigational Product (IP), Within 90 Days After the First IP Administration.
Description: There were no subjects in either treatment group who met the predefined criteria for the primary safety endpoint: the proportion of subjects with TEAEs judged to be probably or definitely related to the IP within 90 days after the first IP administration.
Time Frame: within 90 days after the first IP administration
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | LT3001 Drug Product | Placebo
Number analyzed (Participants) | 43 | 44
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time the subject received the first IP until the last follow-up visit, approximately 92 days.
Description: The same definitions from the clinicaltrials.gov.
Arm/Group | LT3001 Drug Product | Placebo
All-Cause Mortality (participants affected / at risk) | 4/43 | 1/44
Serious Adverse Events (participants affected / at risk) | 12/43 | 5/44
Other Adverse Events (participants affected / at risk) | 37/43 | 33/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LT3001 Drug Product (N=43) | Placebo (N=44)
Stroke, Brain oedema, Encephalopathy, Neurological decompensation (Nervous system disorders) | 6 (6) | 4 (4)
Colitis ischaemic, Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pneumonia, Pneumonia aspiration (Infections and infestations) | 2 (2) | 0 (0)
Fall, Traumatic subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Leukopenia, Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LT3001 Drug Product (N=43) | Placebo (N=44)
Constipation, Diarrhoea (Gastrointestinal disorders) | 17 (32) | 17 (24)
UTI, Pneumonia, Pneumonia aspiration, COVID-19, Conjunctivitis (Infections and infestations) | 18 (27) | 11 (17)
Hyperlipidaemia, Hypokalaemia (Metabolism and nutrition disorders) | 16 (26) | 12 (17)
Headache, Stroke, Brain oedema (Nervous system disorders) | 13 (24) | 9 (13)
Insomnia (Psychiatric disorders) | 9 (9) | 10 (13)
Arthralgia, Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (11) | 7 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 7 (10)
Pyrexia (General disorders) | 6 (8) | 4 (4)
Renal and urinary disorders (Renal and urinary disorders) | 5 (7) | 5 (6)
Cardiac disorders (Cardiac disorders) | 4 (4) | 6 (6)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 6 (8) | 3 (3)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 3 (4) | 5 (5)
Investigations (Investigations) | 1 (1) | 6 (8)
Hypertension (Vascular disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT05403866/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT05403866/SAP_001.pdf